CLINICAL TRIAL: NCT01488708
Title: A Phase 3b, Multicenter, Open-Label Study to Evaluate the Long-Term Safety and Efficacy of Subcutaneous LY2127399 in Participants With Systemic Lupus Erythematosus (SLE) (Illuminate-X)
Brief Title: On Open-Label Study in Participants With Systemic Lupus Erythematosus
Acronym: Illuminate-X
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13811; H9B-MC-BCDX (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Systemic Lupus Erythematosus; Connective Tissue Disease; Autoimmune Disease
Keywords: Lupus; SLE; Systemic Lupus Erythematosus; Immune System Disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases | interventions — tabalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY 2127399 Q2W (Experimental): If participant received LY2127399 in core study: 1 subcutaneous (SC) injection of 120 mg LY2127399 and 1 SC injection of placebo at week 0, followed by 1 SC injection of 120 mg LY2127399 every 2 weeks (Q2W) for 216 weeks. If participant received placebo in core study: 2 SC injections of 120 mg LY2127399 at Week 0, followed by 1 SC injection of 120 mg LY2127399 Q2W for 216 weeks.
  Interventions: Drug: LY2127399; Drug: Placebo
- LY2127399 Q4W (Experimental): If participant received LY2127399 in core study: 1 subcutaneous (SC) injection of 120 mg LY2127399 and 1 SC injection of placebo at Week 0, followed by 1 SC injection of 120 mg LY2127399 every 4 weeks (Q4W) for 216 weeks. If participant received placebo in core study: 2 SC injections of 120 mg LY2127399 at week 0, followed by 1 SC injection of 120 mg LY2127399 Q4W for 216 weeks.
  Interventions: Drug: LY2127399; Drug: Placebo

INTERVENTIONS:
Drug: LY2127399 — 120 mg LY2127399 administered via subcutaneous (SC) injection for 216 weeks Participants randomized to active treatment in the core studies will remain on the same active dose. In order to ensure that the original randomization arm from the preceding core studies is not unblinded, the first dose in BCDX will be blinded, with all participants receiving 2 injections of blinded study drug.
Drug: Placebo — Placebo administered via SC injection at first dose to maintain blinding of previous study treatment.

SUMMARY:
The purpose of this SLE study is to evaluate the long-term safety and efficacy of LY2127399 in eligible SLE participants who have completed the core studies (NCT01196091) (NCT01205438).

ELIGIBILITY:
Inclusion Criteria:

* Have completed 52 weeks of treatment in core studies (NCT01196091) (NCT01205438)
* Given written informed consent
* Test negative for pregnancy at the time of enrollment
* Agree to use a reliable method of birth control

Exclusion Criteria:

* Unwilling to comply with study procedures
* Any condition that renders the participants unable to understand the nature and scope and possible consequences of the study
* Any condition that in the opinion of the investigator poses an unacceptable risk to the participants if study drug would be administered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1518 (Actual)
Dates: Start 2012-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559 or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT-5 hours, EST, Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Irving, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY 2127399 Q2W | LY2127399 Q4W
Started | 940 | 578
Received at Least 1 Dose of Study Drug | 937 | 578
Participated in Follow Up | 810 | 526
Completed | 0 | 0
Not Completed | 940 | 578

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY 2127399 Q2W | LY2127399 Q4W | Total
Number analyzed (Participants) | 940 | 578 | 1518
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (12.12) | 40.4 (11.35) | 42.4 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 880 | 527 | 1407
  Male | 60 | 51 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 265 | 189 | 454
  Not Hispanic or Latino | 612 | 314 | 926
  Unknown or Not Reported | 63 | 75 | 138
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 104 | 94 | 198
  Asian | 113 | 96 | 209
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 130 | 33 | 163
  White | 579 | 337 | 916
  More than one race | 14 | 17 | 31
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 449 | 83 | 532
  Puerto Rico | 14 | 1 | 15
  Canada | 3 | 3 | 6
  Peru | 31 | 38 | 69
  Brazil | 18 | 36 | 54
  Mexico | 23 | 28 | 51
  Ecuador | 21 | 20 | 41
  Argentina | 16 | 23 | 39
  Colombia | 18 | 12 | 30
  Guatemala | 14 | 16 | 30
  Chile | 7 | 3 | 10
  Philippines | 33 | 26 | 59
  Taiwan | 22 | 20 | 42
  Japan | 17 | 19 | 36
  South Korea | 15 | 14 | 29
  Thailand | 14 | 10 | 24
  Australia | 6 | 3 | 9
  New Zealand | 2 | 3 | 5
  Malaysia | 2 | 0 | 2
  Singapore | 0 | 1 | 1
  Serbia | 27 | 36 | 63
  Hungary | 21 | 23 | 44
  Poland | 22 | 19 | 41
  Russia | 17 | 21 | 38
  Ukraine | 14 | 17 | 31
  Romania | 13 | 10 | 23
  Spain | 10 | 12 | 22
  Germany | 11 | 4 | 15
  Belarus | 4 | 7 | 11
  Bulgaria | 7 | 4 | 11
  Latvia | 5 | 4 | 9
  Macedonia | 5 | 3 | 8
  Austria | 1 | 3 | 4
  Italy | 1 | 2 | 3
  Croatia | 1 | 1 | 2
  France | 1 | 1 | 2
  Tunisia | 21 | 19 | 40
  South Africa | 13 | 18 | 31
  Israel | 13 | 9 | 22
  Egypt | 5 | 4 | 9
  United Kingdom | 3 | 2 | 5
Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA-SLEDAI) Score [Mean (Standard Deviation); unit: units on a scale] — SELENA SLEDAI is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105; scores > 20 are rare.
  units on a scale | 5.4 (3.81) | 4.9 (3.74) | 5.2 (3.79)
Anti-dsDNA Antibody Level (IU) [Mean (Standard Deviation); unit: International Unit/Milliliter (IU/mL)] | 82.9 (102.03) | 92.3 (102.35) | 86.4 (102.23)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: Baseline through 4 years
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LY 2127399 Q2W | LY2127399 Q4W
Number analyzed (Participants) | 937 | 578
percentage of participants | 73.3 | 65.6

2. Secondary Outcome: Proportion of Participants With a Systemic Lupus Erythematosus (SLE) Responder Index (SRI) Response
Time Frame: Week 48
Population: Zero participants analyzed. Data was not collected for analysis.
Arm/Group | LY 2127399 Q2W | LY2127399 Q4W
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Proportion of Participants With a Reduction in Steroid Dose
Time Frame: Baseline through 4 years
Population: Zero participants analyzed. Data was not collected for analysis.
Arm/Group | LY 2127399 Q2W | LY2127399 Q4W
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in SLE Disease Activity Index
Time Frame: Baseline, 4 years
Population: Zero participants analyzed. Data was not collected for analysis.
Arm/Group | LY 2127399 Q2W | LY2127399 Q4W
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Occurrence of New Severe SLE Flares
Time Frame: Baseline through 4 years
Population: Zero participants analyzed. Data was not collected for analysis.
Arm/Group | LY 2127399 Q2W | LY2127399 Q4W
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Proportion of Participants With Improvement in Lupus Quality of Life
Time Frame: 4 years
Population: Zero participants analyzed. Data was not collected for analysis.
Arm/Group | LY 2127399 Q2W | LY2127399 Q4W
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Anti-double-stranded Deoxyribonucleic Acid Level
Time Frame: Baseline, 4 years
Population: Zero participants analyzed. Data was not collected for analysis.
Arm/Group | LY 2127399 Q2W | LY2127399 Q4W
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug.
Groups:
- LY 2127399 Q2W Treatment: If participant received LY2127399 in core study: 1 subcutaneous (SC) injection of 120 mg LY2127399 and 1 SC injection of placebo at week 0, followed by 1 SC injection of 120 mg LY2127399 every 2 weeks (Q2W) for 216 weeks. If participant received placebo in core study: 2 SC injections of 120 mg LY2127399 at Week 0, followed by 1 SC injection of 120 mg LY2127399 Q2W for 216 weeks.
  LY2127399: 120 mg LY2127399 administered via subcutaneous (SC) injection for 216 weeks Participants randomized to active treatment in the core studies will remain on the same active dose. In order to ensure that the original randomization arm from the preceding core studies is not unblinded, the first dose in BCDX will be blinded, with all participants receiving 2 injections of blinded study drug.
  Placebo: Placebo administered via SC injection at first dose to maintain blinding of previous study treatment.
- LY2127399 Q4W Treatment: If participant received LY2127399 in core study: 1 subcutaneous (SC) injection of 120 mg LY2127399 and 1 SC injection of placebo at Week 0, followed by 1 SC injection of 120 mg LY2127399 every 4 weeks (Q4W) for 216 weeks. If participant received placebo in core study: 2 SC injections of 120 mg LY2127399 at week 0, followed by 1 SC injection of 120 mg LY2127399 Q4W for 216 weeks.
  LY2127399: 120 mg LY2127399 administered via subcutaneous (SC) injection for 216 weeks Participants randomized to active treatment in the core studies will remain on the same active dose. In order to ensure that the original randomization arm from the preceding core studies is not unblinded, the first dose in BCDX will be blinded, with all participants receiving 2 injections of blinded study drug.
  Placebo: Placebo administered via SC injection at first dose to maintain blinding of previous study treatment.
- LY 2127399 Q2W Follow Up: If participant received LY2127399 in core study: 1 subcutaneous (SC) injection of 120 mg LY2127399 and 1 SC injection of placebo at week 0, followed by 1 SC injection of 120 mg LY2127399 every 2 weeks (Q2W) for 216 weeks. If participant received placebo in core study: 2 SC injections of 120 mg LY2127399 at Week 0, followed by 1 SC injection of 120 mg LY2127399 Q2W for 216 weeks. Follow up.
- LY2127399 Q4W Follow Up: If participant received LY2127399 in core study: 1 subcutaneous (SC) injection of 120 mg LY2127399 and 1 SC injection of placebo at Week 0, followed by 1 SC injection of 120 mg LY2127399 every 4 weeks (Q4W) for 216 weeks. If participant received placebo in core study: 2 SC injections of 120 mg LY2127399 at week 0, followed by 1 SC injection of 120 mg LY2127399 Q4W for 216 weeks. Follow up.
Arm/Group | LY 2127399 Q2W Treatment | LY2127399 Q4W Treatment | LY 2127399 Q2W Follow Up | LY2127399 Q4W Follow Up
Serious Adverse Events (participants affected / at risk) | 129/937 | 64/578 | 57/810 | 51/526
Other Adverse Events (participants affected / at risk) | 464/937 | 232/578 | 37/810 | 24/526
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY 2127399 Q2W Treatment (N=937) | LY2127399 Q4W Treatment (N=578) | LY 2127399 Q2W Follow Up (N=810) | LY2127399 Q4W Follow Up (N=526)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block bilateral (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Tricuspid valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Mineralocorticoid deficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site erosion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Pelvic mass (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amoebiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blastocystis infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Cervicitis (Infections and infestations) | 0/877 (0) | 1/527 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Herpes zoster disseminated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 11 (12) | 1 (1) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 3 (3)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vulval cellulitis (Infections and infestations) | 1/877 (1) | 0/527 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QRS complex shortened (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesterosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 8 (9) | 2 (2) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4) | 1 (1) | 5 (5)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/877 (1) | 0/527 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/877 (1) | 0/527 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0/50 (0) | 1/44 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0/760 (0) | 1/482 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/877 (1) | 0/527 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/877 (1) | 0/527 (0) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery dissection (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IIIrd nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neuropsychiatric lupus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
VIth nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1/877 (1) | 0/527 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/877 (1) | 1/527 (1) | 0 (0) | 0 (0)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0/760 (0) | 1/482 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/877 (1) | 0/527 (0) | 1/760 (1) | 0/482 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium tremens (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (3) | 2 (2) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/60 (0) | 1/51 (1) | 0/50 (0) | 1/44 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/877 (0) | 1/527 (1) | 0/760 (0) | 1/482 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1/877 (1) | 0/527 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/877 (0) | 1/527 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucocutaneous ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 1 (3) | 1 (1) | 1 (1) | 1 (1)
Infarction (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Poor venous access (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY 2127399 Q2W Treatment (N=937) | LY2127399 Q4W Treatment (N=578) | LY 2127399 Q2W Follow Up (N=810) | LY2127399 Q4W Follow Up (N=526)
Abdominal pain (Gastrointestinal disorders) | 21 (21) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9) | 12 (12) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 59 (70) | 18 (21) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 (24) | 7 (7) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 34 (36) | 12 (14) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 21 (23) | 10 (10) | 0 (0) | 0 (0)
Fatigue (General disorders) | 19 (20) | 7 (7) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 20 (25) | 4 (4) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 57 (74) | 26 (32) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 14 (18) | 16 (16) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 63 (83) | 40 (46) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 27 (33) | 15 (16) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 56 (64) | 17 (28) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 104 (142) | 51 (68) | 18 (18) | 11 (12)
Urinary tract infection (Infections and infestations) | 106 (158) | 52 (78) | 20 (21) | 16 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (39) | 12 (16) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (39) | 17 (17) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (29) | 6 (8) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 18 (19) | 12 (13) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 53 (67) | 28 (34) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 21 (21) | 10 (11) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 18 (18) | 12 (12) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (29) | 10 (13) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 23 (28) | 6 (8) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 27 (27) | 8 (10) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated early due to lack of efficacy in parent studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days